CLINICAL TRIAL: NCT03330769
Title: Ultrasound in PSoriatic Arthritis TREAtMent - UPSTREAM
Brief Title: Ultrasound in Psoriatic Arthritis Treatment
Acronym: UPSTREAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Italian Society for Rheumatology (Other); University of Turin, Italy (Other); University Hospital, Udine, Italy (Other); Azienda Sanitaria Locale Roma E (Other)
Responsible Party: Principal Investigator, Matteo Piga, Researcher, University of Cagliari
Other Study IDs: F8MRG
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Arthritis, Psoriatic; Ultrasonography; Minimal Disease, Residual
Keywords: Psoriatic Arthritis; Ultrasonography; Minimal disease activity
MeSH Terms: conditions — Arthritis, Psoriatic; Neoplasm, Residual | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with active Psoriatic Arthritis: Patients with clinically diagnosed PsA with clinically active joint disease starting a new course of treatment.
  Interventions: Drug: New course of treatment

INTERVENTIONS:
Drug: New course of treatment — Prescription of new course of NSAIDs (monotherapy), steroid intra-articular injections (monotherapy), conventional DMARDs, biologic DMARDs, including switches or dose augmentations, indicated by the treating rheumatologist according to usual clinical practice.
  Other Names: NSAIDs; steroid intra-articular injections; Conventional DMARDs; biologic DMARDs

SUMMARY:
BACKGROUND Psoriatic arthritis (PsA) is a systemic inflammatory disease with articular and extra-articular features. Establishing the prognosis of a patient with PsA is hence important to define the treatment strategy. Currently, observational and prospective cohort studies have identified prognostic factors correlating with the achievement of therapeutic response. Nevertheless, despite the importance of identifying prognostic factors in a disease with a functional disability comparable to rheumatoid arthritis, the studies are still limited.

PRIMARY OBJECTIVE In PsA with clinically active joint disease starting a new course of therapy, to evaluate the additional value of UltraSound(US)-score over clinical examination in detecting patients achieving MDA at 6 months.

STUDY DESIGN The study follows a multi-centre observational prospective cohort study design.

PATIENTS AND METHODS INCLUSION CRITERIA

* Adult > 18 years of age with PsA (PsA according to the ClASsification criteria for Psoriatic Arthritis (CASPAR) - with joint involvement)
* At least one joint clinically involved (both swelling and tenderness);
* prescription of new course of d NSAIDs (monotherapy), steroid intra-articular injections (monotherapy), conventional Disease-Modifying AntiRheumatic Drugs (DMARDs), biologic DMARDs, including switches or dose augmentations indicated by the treating rheumatologist according to usual clinical practice before US acquisition;
* Stable treatment before treatment modification (6 weeks);
* Signed informed consent form.

CLINICAL ASSESSMENT Patient's clinical assessment will be performed according to the core set of domains for PsA proposed by the Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) and Outcome Measures in Rheumatology (OMERACT).

ULTRASOUND ASSESSMENT Sonographic evaluations will be performed by expert ultrasonographers in 44 joints, 36 tendons, 12 entheses and 2 bursae according to the score developed for psoriatic arthritis by the study group ultrasound of the Italian Society of Rheumatology (US-score PsA-SIR)

EXPECTED RESULTS AND SIGNIFICANCE The aim of this study is to identify clinical and US predictors of achieving MDA in PsA patients with active peripheral arthritis starting a new course of therapy.

DETAILED DESCRIPTION:
BACKGROUND Psoriatic arthritis (PsA) is a systemic inflammatory disease with articular and extra-articular features. To date remission is considered to be the ultimate goal of therapy in PsA, however, due to the characteristics of the disease with involvement of different domains, remission may be difficult to achieve and maintain and so a minimal disease activity (MDA) could be an acceptable goal. In view of the therapeutic target of remission or MDA, the identification of adverse prognostic factors and the best treatment strategy are two of the most important items in research agenda of PsA. Establishing the prognosis of a patient with PsA is hence important to define the treatment strategy. Currently, observational and prospective cohort studies have identified prognostic factors correlating with the achievement of therapeutic response. Nevertheless, despite the importance of identifying prognostic factors in a disease with a functional disability comparable to rheumatoid arthritis (RA), the studies are still limited. Undoubtedly, the concept of treat-to-target (T2T) in PsA needs further studies, especially with longer follow up and larger samples. In T2T strategies, it is necessary to quantify the disease activity and this is possible by composite indices. The heterogeneity of PsA including axial and peripheral involvement and specific features (i.e. dactylitis, enthesitis) as well as extra-articular features makes the use of a single composite index (e.g. Disease Activity for Psoriatic Arthritis-DAPSA, Composite Psoriatic Disease Activity Index-CPDAI) a challenge not resolved yet. An interesting possibility is to integrate musculoskeletal ultrasonography (US) with clinical examination to stratify patients and to decide treatments in a T2T strategy. In the last years the role of imaging is grown up and EULAR recommendations on the use of imaging techniques in chronic arthritis recognize the high sensitivity of US to detect disease activity better than clinical examination alone although the utility of US in clinical practice is not supported by sufficient evidence yet

AIM

The aim of this study is to identify clinical and US predictors of achieving MDA in PsA patients with active peripheral arthritis starting a new course of therapy.

Identifying prognostic factors of achieving remission or low disease activity will allow a better selection of patients with poorer outcome and a following improvement of the therapeutic strategies. Furthermore the possibility that US could be an added prognostic value makes this study a clear example of integration between the clinic and US. This study will respond to the need of tailoring treatment that would allow clinicians to practice a more effective and personalized medicine, optimizing the outcomes of patients with PsA as well as the treatments management.

STUDY OBJECTIVES

PRIMARY OBJECTIVE

In clinically diagnosed PsA with clinically active joint disease starting a new course of therapy, to evaluate the additional value of US-score (US-score PsA-SIR) over clinical examination in detecting patients achieving MDA at 6 months.

SECONDARY OBJECTIVES

In clinically diagnosed PsA with clinically active joint disease starting a new course of therapy:

* to evaluate the additional value of US over clinical examination in detecting patients:
* achieving MDA at 12 months (including sustained)
* achieving DAPSA remission at 6 and 12-months (including sustained)
* achieving American College of Rheumatology (ACR) remission at 6 and 12 months (including sustained)
* with X-ray structural progression using the modified Sharp-van der Heijde score (mSvHs) at 12 and 24 months
* with US structural progression (US-damage score) at 12 and 24 months
* with functional worsening measured using Health Assessment Questionnaire (delta HAQ>0.23) at 12 and 24 months
* with impairment of Health Related Quality of Life (HRQoL) measured with Psoriatic Arthritis Impact of Disease (PsAID) questionnaire at 12 and 24 months;
* to evaluate the relationship between time-integrated US-detected inflammation and US-detected damage at 12 and 24 months;
* to evaluate the comparative effectiveness of different treatment strategies on MDA, DAPSA remission, HAQ>0.23, X-ray progression (mSvHs), US-inflammation score, US-damage score;
* to evaluate residual US activity in patients in MDA remission;
* to explore whether clinically-detected disease activity due to joint tenderness without swelling is related to joint or extra-articular US-detected inflammation evaluated by US;
* to explore clinical features and US-lesions related to X-ray detected bony apposition.

STUDY DESIGN

The study follows a multi-centre observational prospective cohort study design.

SAFETY MONITORING

An adverse event (AE) is any untoward medical occurrence (i.e., any unfavourable and unintended sign (including abnormal laboratory findings), symptom or disease) in a subject after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a specific medicinal product.

DEFINITION OF SAE

An SAE is defined as any adverse event (appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s) or medical conditions(s) which meets any one of the following criteria:

* is fatal or life-threatening
* results in persistent or significant disability/incapacity
* constitutes a congenital anomaly/birth defect
* requires inpatient hospitalization or prolongation of existing hospitalization.

STATISTICAL ANALYSIS PLAN VARIABLES

OUTCOME MEASURES

PRIMARY:

o MDA at 6 months

SECONDARY:

* MDA at 12 months, sustained MDA at 6 AND 12 months
* DAPSA <3.3 at 6 months, 12 months, 6 AND 12 months
* deltam SvHs 0-12 and 0-24 months
* delta HAQ 0-12 and 0-24 months
* delta PSAID 0-12 and 0-24 months
* US-score PsA-SIR damage subscore at 0-6-12 months US PREDICTORS
* US-score PsA-SIR
* US-score PsA-SIR inflammation subscore
* US-score PsA-SIR damage subscore

CLINICAL PREDICTORS

Based on the relevant literature clinical variables to be considered in the model include:

* Demographic and environmental factors:
* Age
* Gender
* Smoking
* BMI
* Clinical factors:
* subset of PsA
* time from symptoms onset to diagnosis
* disease duration
* disease activity (DAPSA and BASDAI)
* HAQ score
* tender joints / pain
* comorbidities (FM, MetS)
* Serological factors:
* Acute phase reactants
* Therapy factors:
* Treatment (NSAIDs, steroids, DMARDs)

DESCRIPTIVE ANALYSES

Descriptive data will be provided for all outcomes according to data type; number of patients (N), mean, standard deviation (for interval data), median 25% and 75% quartiles (for ordinal data). Frequency (absolute and relative) distributions will be provided for categorical data. Two-sided p-values will be presented throughout.

PRIMARY ENDPOINT ANALYSIS

Prediction of 6 month MDA will use multivariate adjusted logistic models. A baseline model will include all the clinical variables. US predictors will be added as covariates to the clinical variables, assuming an additive model. The derived ß coefficients were used to calculate prognostic indices, thereby creating weighted prediction models.

Model performance will be evaluated by C-indices (area under the ROC curve, AUC), net reclassification indices (NRI), integrated discrimination improvement (IDI), and plotted ROC curves. NRI can be used to compare the clinical impact of different models (it is a comparison of the proportion of subjects with disease who have appropriately increased risk scores with the new model, and the proportion of subjects without disease who have appropriately decreased risk scores with the new model). IDI represents desired improvements in average sensitivity corrected for undesirable increases in 1-specificity, it therefore compared whether the new models improved sensitivity without affecting specificity.( ) Data management and analysis will be performed using RedCap, R, Stata.

SAMPLE SIZE

The sample size calculation was done with the objective of minimizing the number of false positives (i.e the number of false non-responsive to treatment) in order to minimize the risk of over-treating patients who actually have a good response to therapy. Therefore, sample size was calculated to minimize this risk by 40% (null hypothesis H0) to 20% (alternative hypothesis H1), maintaining stable at 70% (both for the H0 for both the H1), the percentage of true positives (true unresponsive to therapy).

The simulations were carried out using the procedure rocsize Stata (by M. Pepe) 30, which allows to determine the power to detect an improvement in the ROC curve. The procedure requires the specification of the percentage of false positive and true positive both for the null hypothesis is for the alternative hypothesis and the percentage of positive / diseased.

Using the command rocsize 0.7 0.2, na (150) ndb (100) tpnull (0.7) fpnull (0.4) of Stata, 250 patients are sufficient to evaluate the performance of a model (and its ROC curve) with 90% power and 5% alpha. Specifically, we have assumed a 70% and a 20% of subjects true positives and false positives, respectively, according to the alternative hypothesis, a 70% and a 40% of subjects true positives and false positives, respectively, according to the null hypothesis, and a percentage of diseased of 60% (150 of 250 subjects).

Under the assumption of maximum attrition of 20%, the sample size will be increased to 300 patients. The same sample size is sufficient to precisely estimate a logistic model of achievement of a MDA (probability of 0.4 at 6 months) with 10 predictors (rule of thumbs).( ) Based on the pre-study activities, 35-40 centres will be involved, 15 tertiary and 20-25 secondary rheumatology centres. Assuming 4 eligible patients/months for tertiary and 1/month in secondary centres, a 40% of enrolment rate, about 30 patients/months are expected.

ETHICS

This study will be conducted in accordance with all applicable laws and regulations including, but not limited to, the International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP), EU guidelines and the ethical principles that have their origins in the Declaration of Helsinki. The institutional review board (IRB)/independent ethics committee (IEC) must review and approve the protocol and informed consent form before any subjects are enrolled. Before any protocol-required procedures are performed, the subject must sign and date the IRB/IEC-approved informed consent form.

Clinical data (including AEs and concomitant medications) will be entered into a validated data capture system provided by the Italian Society for Rheumatology. The data system will include password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years of age with PsA (according to the CASPAR classification Criteria)

  * Clinically active arthritis, with at least one joint clinically involved (both swelling and tenderness) in patient not achieving the MDA;
  * Subject newly prescribed NSAIDs (monotherapy), steroid intra-articular injections (monotherapy), conventional DMARD, biologic DMARDs as indicated by the treating rheumatologist according to usual clinical practice before US acquisition;
  * Stable treatment before treatment modification (6 weeks);
  * Signed informed consent form;

Exclusion Criteria:

* Minimal disease activity a the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically diagnosed PsA with clinically active joint disease starting a new course of therapy for active joint disease.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-29 (Estimated)

PRIMARY OUTCOMES:
Minimal disease activity | 6 months
  The Minimal disease activity (MDA) calculation will be based on the evaluation of 7 variables:
  1. 68 tender joints count (≤1)
  2. 66 swollen joint count (≤1)
  3. Body Surface Area (BSA) ≤3
  4. Patient pain VAS (≤15 mm);
  5. Patient global disease activity VAS (≤20 mm);
  6. HAQ (≤0.5);
  7. Leeds Enthesitis Index (LEI) tender entheseal points (≤1) Patients will be classified as having MDA if they meet 5 out of these 7 criteria (value in brackets).

SECONDARY OUTCOMES:
Minimal disease activity | 12 months
  The Minimal disease activity (MDA) calculation will be based on the evaluation of 7 variables:
  1. 68 tender joints count (≤1)
  2. 66 swollen joint count (≤1)
  3. BSA ≤3
  4. Patient pain VAS (≤15 mm);
  5. Patient global disease activity VAS (≤20 mm);
  6. HAQ (≤0.5);
  7. Leeds Enthesitis Index (LEI) tender entheseal points (≤1)
  Patients will be classified as having MDA if they meet 5 out of these 7 criteria (value in brackets).
Disease Activity for Psoriatic Arthritis (DAPSA) | 6 and 12 months
  The DAPSA calculation is based on the evaluation of 5 variables:
  1. 68 tender joints count (TJC)
  2. 66 swollen joint count (SJC)
  3. Patient's pain (VAS)
  4. Patient's global disease activity assessment (VAS)
  5. C-reactive protein
  As a result the DAPSA index gives a value with:
  >28 indicating high disease activity 14-28 indicating moderate disease activity 4-13 indicating low disease activity
  ≤4 indicating complete remission
  Using DAPSA the clinical response can be defined:
  Minor : 50% DAPSA change from baseline Moderate: 75% DAPSA change from baseline Major : 85% DAPSA change from baseline
American College of Rheumatology (ACR) response score | 6 and 12 months
  The ACR 20 response criteria require ≥ 20% [ACR 50 ≥ 50% or ACR 70 ≥ 70%] improvement in both the TJC and SJC, as well as a 20% improvement in 3 of the following 5 items:
  1. patient global assessments of disease activity (VAS),
  2. patient reported pain score (VAS),
  3. physician global assessment (VAS),
  4. Health Assessment Questionnaire (HAQ),
  5. either Erythrocyte Sedimentation Rate (ESR) or C-Reactive Protein (CRP).
X-ray structural progression (mSVH score) | 12 and 24 months
  Using the modified Sharp-Vander Heijde score. at 12 and 24 months
Ultraosund structural progression | 12 and 24 months
  US-damage score
Functional worsening | 12 and 24 months
  Functional worsening with a delta HAQ>0.23.
Health Related Quality of life | 12 and 24 months
  Impairment of HRQoL using the PSAID-12 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Iagnocco, Prof, Principal Investigator — Università di Torino, Italy; Alen Zabotti, MD, Principal Investigator — University Hospital "Santa Maria della Misericordia", Udine, Italy; Marco Canzoni, Principal Investigator — Local Health Unit (ASL) Rome-1, Rome-4, Viterbo, Italy; Ignazio Benedetto Olivieri, Study Chair — Italian Society of Rheumatology
Locations (4):
- Italy (4):
  - Azienda Ospedaliera Universitaria, Cagliari
  - Local Health Unit (ASL) Rome-1, Rome-4, Roma
  - University of Turin, Torino
  - University Hospital "Santa Maria della Misericordia", Udine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available to all investigators participating in the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 12 months of study completion.
Access Criteria: Data access requests will be reviewed by the Steering Committee and by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Moll JM, Wright V. Psoriatic arthritis. Semin Arthritis Rheum. 1973;3(1):55-78. doi: 10.1016/0049-0172(73)90035-8. No abstract available. PMID 4581554
- [Background] Coates LC, Helliwell PS. Validation of minimal disease activity criteria for psoriatic arthritis using interventional trial data. Arthritis Care Res (Hoboken). 2010 Jul;62(7):965-9. doi: 10.1002/acr.20155. PMID 20589696
- [Background] Gossec L, Smolen JS, Ramiro S, de Wit M, Cutolo M, Dougados M, Emery P, Landewe R, Oliver S, Aletaha D, Betteridge N, Braun J, Burmester G, Canete JD, Damjanov N, FitzGerald O, Haglund E, Helliwell P, Kvien TK, Lories R, Luger T, Maccarone M, Marzo-Ortega H, McGonagle D, McInnes IB, Olivieri I, Pavelka K, Schett G, Sieper J, van den Bosch F, Veale DJ, Wollenhaupt J, Zink A, van der Heijde D. European League Against Rheumatism (EULAR) recommendations for the management of psoriatic arthritis with pharmacological therapies: 2015 update. Ann Rheum Dis. 2016 Mar;75(3):499-510. doi: 10.1136/annrheumdis-2015-208337. Epub 2015 Dec 7. PMID 26644232
- [Background] Saber TP, Ng CT, Renard G, Lynch BM, Pontifex E, Walsh CA, Grier A, Molloy M, Bresnihan B, Fitzgerald O, Fearon U, Veale DJ. Remission in psoriatic arthritis: is it possible and how can it be predicted? Arthritis Res Ther. 2010;12(3):R94. doi: 10.1186/ar3021. Epub 2010 May 18. PMID 20482783
- [Background] Glintborg B, Ostergaard M, Krogh NS, Andersen MD, Tarp U, Loft AG, Lindegaard HM, Holland-Fischer M, Nordin H, Jensen DV, Olsen CH, Hetland ML. Clinical response, drug survival, and predictors thereof among 548 patients with psoriatic arthritis who switched tumor necrosis factor alpha inhibitor therapy: results from the Danish Nationwide DANBIO Registry. Arthritis Rheum. 2013 May;65(5):1213-23. doi: 10.1002/art.37876. PMID 23460467
- [Background] Coates LC, Moverley AR, McParland L, Brown S, Navarro-Coy N, O'Dwyer JL, Meads DM, Emery P, Conaghan PG, Helliwell PS. Effect of tight control of inflammation in early psoriatic arthritis (TICOPA): a UK multicentre, open-label, randomised controlled trial. Lancet. 2015 Dec 19;386(10012):2489-98. doi: 10.1016/S0140-6736(15)00347-5. Epub 2015 Oct 1. PMID 26433318
- [Background] Mandl P, Navarro-Compan V, Terslev L, Aegerter P, van der Heijde D, D'Agostino MA, Baraliakos X, Pedersen SJ, Jurik AG, Naredo E, Schueller-Weidekamm C, Weber U, Wick MC, Bakker PA, Filippucci E, Conaghan PG, Rudwaleit M, Schett G, Sieper J, Tarp S, Marzo-Ortega H, Ostergaard M; European League Against Rheumatism (EULAR). EULAR recommendations for the use of imaging in the diagnosis and management of spondyloarthritis in clinical practice. Ann Rheum Dis. 2015 Jul;74(7):1327-39. doi: 10.1136/annrheumdis-2014-206971. Epub 2015 Apr 2. PMID 25837448
- [Background] Gladman DD, Mease PJ, Healy P, Helliwell PS, Fitzgerald O, Cauli A, Lubrano E, Krueger GG, van der Heijde D, Veale DJ, Kavanaugh A, Nash P, Ritchlin C, Taylor W, Strand V. Outcome measures in psoriatic arthritis. J Rheumatol. 2007 May;34(5):1159-66. PMID 17477479
- [Background] Gladman DD, Mease PJ, Strand V, Healy P, Helliwell PS, Fitzgerald O, Gottlieb AB, Krueger GG, Nash P, Ritchlin CT, Taylor W, Adebajo A, Braun J, Cauli A, Carneiro S, Choy E, Dijkmans B, Espinoza L, van der Heijde D, Husni E, Lubrano E, McGonagle D, Qureshi A, Soriano ER, Zochling J. Consensus on a core set of domains for psoriatic arthritis. J Rheumatol. 2007 May;34(5):1167-70. PMID 17477480
- [Derived] Canzoni M, Piga M, Zabotti A, Scire CA, Carrara G, Olivieri I, Iagnocco A. Clinical and ultrasonographic predictors for achieving minimal disease activity in patients with psoriatic arthritis: the UPSTREAM (Ultrasound in PSoriatic arthritis TREAtMent) prospective observational study protocol. BMJ Open. 2018 Jul 10;8(7):e021942. doi: 10.1136/bmjopen-2018-021942. PMID 29991631

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03330769/Prot_SAP_000.pdf